CLINICAL TRIAL: NCT00172757
Title: Risk Factors of Colorectal Cancer in Taiwan-With Special Reference to the Association With Nutrition, Diet, Obesity, Diabetes Mellitus, and Genetic Alterations
Brief Title: Association of Colorectal Cancer With Nutrition, Diet, Obesity, Diabetes Mellitus, and Genetic Alterations in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701298
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-11-28 (Estimated); Status verified 2003-01

CONDITIONS: Colorectal Cancer
Keywords: MSI, TS, Colorectal Cancer, DM.
MeSH Terms: conditions — Colorectal Neoplasms; Microsatellite Instability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
We will explore the genetic (including APC, k-ras, p53, MSI, etc.) and environmental (including family history, life style, diet, nutritional status, DM, serum IGF-I, IGFBP-3, etc.) risk factors of colorectal tumorigenesis. We will accrue approximately 1000 patients as experimental group. The control group consists of 2000 individuals who were confirmed without colorectal cancer or polyps by colonoscopy. We estimated the statistical power of this study will reach more than 90%. In the second year, we will explore the association between various environmental risk factors with the epigenetic changes of various oncogenes and tumor suppressor genes. Firstly, we will study the correlation between hypermethylation of promoter region of hMLH1 gene with various environmental factors. Next, we will explore the genetic polymorphisms of promoter of E-cadherin gene. Recently, it has been reported that the C→A genetic polymorphism in the promoter region of E-cadherin gene in prostate cancer. Since this phenomenon has not been reported in colorectal cancer, it is mandatory for us to extend our research to the E-cadherin polymorphisms of colorectal cancer. Moreover, this project will focus on exploration of the association between the genetic polymorphisms of promoter of TS gene with chemosensitivity to 5-Fu-based therapy. We speculated that the better prognosis in colorectal tumors with MSI is related to their expression of TS gene. In summary, the second year of this project will extend our accumulated experience in the study of genetic polymorphisms to further clarify the association between genetic polymorphisms of TS gene with the prognosis of colorectal cancers after chemotherapy. We believe that this project will facilitate: (1) the further clarification of colorectal cancer tumorigenesis; (2) the establishment of domestic epidemiological data of colorectal cancer of Taiwan, and (3) the improvement of the quality of clinical management of patients with colorectal cancer.

DETAILED DESCRIPTION:
This is a two-year hospital-based case control study. In the fist year, we will set up solid database of our laboratory regarding the molecular genetics of colorectal cancer. We will explore the genetic (including APC, k-ras, p53, MSI, etc.) and environmental (including family history, life style, diet, nutritional status, DM, serum IGF-I, IGFBP-3, etc.) risk factors of colorectal tumorigenesis. During the whole 2-year period of this project, we will accrue approximately 1000 patients as experimental group. The control group consists of 2000 individuals who were confirmed without colorectal cancer or polyps by colonoscopy. We estimated the statistical power of this study will reach more than 90%. In the second year, we will explore the association between various environmental risk factors with the epigenetic changes of various oncogenes and tumor suppressor genes. It has been well known that epigenetic changes of various oncogene and tumor suppressor genes was related to the intrinsic and extrinsic environmental alterations. Firstly, we will study the correlation between hypermethylation of promoter region of hMLH1 gene with various environmental factors. Next, we will explore the genetic polymorphisms of promoter of E-cadherin gene. It has been well known that E-cadherin plays a major role in the maintenance of cellular structure. Recently, it has been reported that the C→A genetic polymorphism in the promoter region of E-cadherin gene in prostate cancer. The experimental method was feasible in our laboratory. Since this phenomenon has not been reported in colorectal cancer, it is mandatory for us to extend our research to the E-cadherin polymorphisms of colorectal cancer. Moreover, this project will focus on exploration of the association between the genetic polymorphisms of promoter of TS gene with chemosensitivity to 5-Fu-based therapy. Recent reports indicated that colorectal tumors with MSI have better prognosis. Moreover, some authors indicated that the genetic polymorphisms of TS genes was related to chemosensitivity. Therefore, we speculated that the better prognosis in colorectal tumors with MSI is related to their expression of TS gene. In summary, the second year of this project will extend our accumulated experience in the study of genetic polymorphisms to further clarify the association between genetic polymorphisms of TS gene with the prognosis of colorectal cancers after chemotherapy. We believe that this project will facilitate: (1) the further clarification of colorectal cancer tumorigenesis; (2) the establishment of domestic epidemiological data of colorectal cancer of Taiwan, and (3) the improvement of the quality of clinical management of patients with colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive cases of sporadic colorectal cancer in NTUH.

Exclusion Criteria:

* FAP and HNPCC.

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000
Dates: Start 2002-01; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tung Liang, M.D., Ph.D., Principal Investigator — Department of Surgery, National Taiwan University Hospital, No.7, Chung-Shan South Road, Taipei, TAIWAN, R.O.C.
Locations (1):
- Department of Surgery, National Taiwan University Hospital, No.7, Chung-Shan South Road, Taipei, TAIWAN, R.O.C., Taipei, Taiwan